CLINICAL TRIAL: NCT06642779
Title: Comparative Analysis of the Visual Performance and Patient Satisfaction After Cataract Surgery With Implantation of a Medicontur Monofocal (877PAY) or a Medicontur Extended Depth of Focus (877PEY) IOL
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M_877PAY_877PEY_HU_2020
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cataract; Presbyopia; Ametropia
Keywords: Intraocular lens; monofocal IOL; EDOF
MeSH Terms: conditions — Cataract; Presbyopia; Refractive Errors | interventions — Slit Lamp Microscopy; Ophthalmoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 877PAY (monofocal): 26 patients (52 eyes) binocularly implanted with the 877PAY monofocal IOL model
  Interventions: Behavioral: VFQ- 25 (Visual Function Questionnaire); Diagnostic Test: Optical Biometry; Diagnostic Test: Slit lamps / Fundoscopy / Biomicroscopy; Diagnostic Test: UDVA; Diagnostic Test: CDVA; Diagnostic Test: UIVA / DCIVA; Diagnostic Test: UNVA / DCNVA; Diagnostic Test: Manifest Refraction; Diagnostic Test: IOP; Diagnostic Test: VADC; Diagnostic Test: CSDC; Diagnostic Test: CSV-1000; Diagnostic Test: Tear film stability; Device: IOL implantation
- 877PEY (extended depth of focus): 38 patients (76 eyes) binocularly implanted with the 877PEY extended depth of focus IOL model
  Interventions: Behavioral: VFQ- 25 (Visual Function Questionnaire); Diagnostic Test: Optical Biometry; Diagnostic Test: Slit lamps / Fundoscopy / Biomicroscopy; Diagnostic Test: UDVA; Diagnostic Test: CDVA; Diagnostic Test: UIVA / DCIVA; Diagnostic Test: UNVA / DCNVA; Diagnostic Test: Manifest Refraction; Diagnostic Test: IOP; Diagnostic Test: VADC; Diagnostic Test: CSDC; Diagnostic Test: CSV-1000; Diagnostic Test: Tear film stability; Device: IOL implantation

INTERVENTIONS:
Behavioral: VFQ- 25 (Visual Function Questionnaire) — VFQ-25 questionnaire was used to evaluate patient satisfaction at the M3 and M12 visits.
Diagnostic Test: Optical Biometry — Axial length, anterior chamber depth and corneal keratometric values K1-K2. All these parameters were measured at the screening visit and at the month 3 follow-up visit, using the ARGOS® Biometer or the ANTERION® Cataract App
Diagnostic Test: Slit lamps / Fundoscopy / Biomicroscopy — The fundus and other ocular structures, such as the cornea, anterior chamber, iris, pupil, crystalline lens / IOL alignment, corpus ciliare and choroid were examined at screening visit, on the day of the surgery, and at the follow up visits D1, M1, M3, M6, and M12, using the slit lamp binocular indirect ophthalmoscopy.
Diagnostic Test: UDVA — Monocular and binocular Uncorrected Distance Visual Acuity (UDVA) was evaluated at all visits (preoperative, D1, M1, M3, M6 and M12), using the ETDRS chart.
Diagnostic Test: CDVA — Monocular and binocular Corrected Distance Visual Acuity (UDVA) was evaluated at all visits (preoperative, D1, M1, M3, M6 and M12), using the ETDRS chart.
Diagnostic Test: UIVA / DCIVA — Uncorrected and Distance Corrected Intermediate Visual acuity (UIVA / DCIVA) was evaluated postoperatively at M1, M3, M6 and M12, using an intermediate chart from 67 cm.
Diagnostic Test: UNVA / DCNVA — Uncorrected and Distance Corrected Near Visual acuity (UNVA / DCNVA) was evaluated postoperatively at M1, M3, M6 and M12, using a near chart from 40 cm.
Diagnostic Test: Manifest Refraction — Manifest refraction was the monocular subjective refraction (Sph, Cyl, Axis) giving the best distance corrected visual acuity. It was measured at the screening visit and the follow-up visits Day 1, Month 1, Month 3, Month 6 and Month 12.
Diagnostic Test: IOP — Intraocular pressure (IOP) was measured at all visits (preoperative, D1, M1, M3, M6 and M12), using a non-contact tonometer.
Diagnostic Test: VADC — Visual Acuity Defocus Curve (VADC) was taken monocularly at M3, monocularly and binocularly at M6 and binocularly at M12, using the Multifocal Lens analyzer - MLA application.
Diagnostic Test: CSDC — Contrast Sinsitivity Defocus Curve (CSDC) was taken under photopic conditions at M6 and M12, using the Multifocal Lens Analyzer - MLA application
Diagnostic Test: CSV-1000 — Contrast Sensitivity was measured using the CSV-1000 with distance correction in place at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd). Measurements were taken under four different light conditions:
  * Photopic (M3 monocular and binocular, M6 binocular and M12 monocular)
  * Mesopic (M6 binocular)
  * Photopic with backlight (M6 binocular)
  * Mesopic with backlight (M6 binocular)
Diagnostic Test: Tear film stability — Tear film stability was assessed at screening visit and at follow-up visits M1, M3, M6, and M12 using the non-invasive Tear break Up Time (TBUT) with fluorescein dye.
Device: IOL implantation — The investigational device (877PEY) and the comparator (877PAY) intraocular lens models were implanted, using sutureless, small-incision phacoemulsification surgery.

SUMMARY:
The purpose of this multi-center, prospective, randomized, comparative clinical investigation was to evaluate and compare the visual performance at far, intermediate and near distances, the presence of photopic phenomena and patient satisfaction after cataract surgery in patients implanted binocularly with a Medicontur monofocal (877PAY) or a Medicontur extended depth of focus (877PEY) IOL models.

The visit schedule included a total of 6 visits, in addition to the IOL implantation surgery, with the listed follow-up timeline:

* screening and baseline assessments
* day 0 (IOL implantation surgery)
* day 1
* month 1
* month 3
* month 6
* month 12

ELIGIBILITY:
Inclusion Criteria:

* cataractous patients who wish to be partly spectacle independent
* cataractous lens changes as demonstrated by best corrected visual acuity of 20/40 or worse either with or without a glare source present (e.g., Brightness Acuity Tester) or with significant cataract-related visual symptoms*
* best corrected visual acuity to be better than 20/25 (0.1 logMAR) after cataract removal and IOL implantation*
* ≤ 1.0 D of preoperative keratometric astigmatism;
* clear intraocular media other than cataract;
* given written informed consent by subject;
* subjects are willing and able to comply with schedule for follow-up visits;
* adult patient

Exclusion Criteria:

* corneal astigmatism > 1.00 D
* irregular astigmatism
* diabetic retinopathy
* iris neovascularisation
* serious intraoperative complications
* congenital eye abnormality
* uncontrolled glaucoma or glaucoma with changes in optical nerve and visual field
* pseudoexfoliation syndrome
* amblyopia
* uveitis
* long-term anti-inflammatory treatment
* AMD
* retinal detachment
* prior ocular surgery in personal medical history
* corneal diseases
* severe retinal diseases (dystrophy, degeneration)
* severe myopia (if required IOL power is lower than 10 D)
* inadequate visualization of the fundus on preoperative examination
* patients deemed by the clinical investigator because of any systemic disease.
* eye trauma in medical history

Intraoperative exclusion criteria:

* tear in capsulorhexis*
* zonular dehiscence*
* posterior capsular rupture vitreous loss and other unexpected surgical complication*

  * According to coordinator investigator's decision, the marked inclusion and exclusion criteria were not applied.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (18 years old and older) with cataract and/or ametropia (hyperopia, myopia), who hace signed the informed consent form and undergone binocular implantation with the investigational device (877PEY) or the comparator device (877PAY).
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
DCIVA | measured at month 1, month 3, month 6 and month 12
  distance corrected intermediate visual acuity

SECONDARY OUTCOMES:
UDVA/CDVA | measured at month 1, month 3, month 6 and month 12
  uncorrected and corrected distance visual acuity
VADC | measured at month 3, month 6 and month 12
  visual acuity defocus curves
CSDC | measured at month 6 and month 12
  contrast sensitivity defocus curves
Patient satisfaction | Evaluated at month 3 and month 12
  presence of visual disturbances (glares, halos), evaluated with the VFQ-25 questionnaire.
CSV-1000 | measured at month 3, month 6 and month 12
  Contrast sensitivity measured with the CSV-1000 standardized auto-calibrating vision testing instrument

OTHER OUTCOMES:
Safety (intraoperative complications of cataract surgery) | Up to day 1 postoperatively
  * Posterior capsular or zonular rupture
  * Vitreous loss/anterior vitrectomy or aspiration
  * Iris/ciliary body injury
  * Loss of nuclear material into vitreous
  * Suprachoroidal haemorrhage
  * Retrobulbar hemorrhage
Safety (postoperative complications of cataract surgery) | Up to month 1 postoperatively
  * Cystoid macular edema
  * Iris abnormalities
  * Corneal edema
  * Wound leak or rupture
  * IOL dislocation, removal, or exchange
  * Inflammation (Endophthalmitis, anterior chamber cells, anterior chamber flare, hypopyon)
  * Retinal tear, break, or detachment
  * Persistent iritis
  * Elevated intraocular pressure
  * Pupillary block
  * Cornea status
Safety (complications of IOL implantation) | Up to month 12 postoperatively
  * Posterior capsular opacification (PCO)
  * Opacification, IOL discoloration

CONTACTS AND LOCATIONS:
Overall Officials: József F Győry, MD, Principal Investigator — Retinaszerviz Kft. (8200 Veszprém, Vörösmarty tér 6, Hungary)
Locations (3):
- Hungary (3):
  - Borsod-Abaúj-Zemplén Vármegyei Központi Kórház és Egyetemi Oktatókórház, Miskolc, BAZ Vármegye
  - Győr-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Győr, Győr-Moson-Sopron Vármegye
  - Retinaszerviz Kft., Veszprém, Veszprém Vármegye